CLINICAL TRIAL: NCT04106154
Title: Impacting Children's Physical and Mental Health Through Kinesiology Support in Clinical Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Pat Longmuir, Senior Scientist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19/115X
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Congenital Heart Defect; Chronic Pain; Concussion Post Syndrome; Cerebral Palsy; Neuromuscular Diseases; Physical Disability
Keywords: Physical Activity; Activity Motivation; Activity Confidence; Children; Adolescents; Sleep; Screen Time
MeSH Terms: conditions — Heart Defects, Congenital; Chronic Pain; Post-Concussion Syndrome; Cerebral Palsy; Neuromuscular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A research assistant or graduate student blind to participants' intervention status will complete all measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The kinesiology intervention will involve physical activity education appropriate to the MC&D delivered in a group format through twelve 2.5-hour weekly sessions49 (30 hours of kinesiology support). The sessions will combine participation in physical activities appropriate to the MC&D with education and goal-setting discussions. Each week, children will be guided to develop an individualized SMART (Specific, Measurable, Agreed upon, Realistic, Time-based) plan for changing their activity behaviour. Their weekly SMART plan, which will require an additional 2 hours per week, will specify the home/community activities they will do prior to the next session.
  Interventions: Behavioral: Kinesiology Support
- Control (No Intervention): Patients in the control group will continue with clinical care as usual. To encourage their cooperation, children in the control group will be offered the intervention after all of their study visits have been completed.

INTERVENTIONS:
Behavioral: Kinesiology Support — 12 week physical activity group led by Kinesiologist. The intervention will be used to increase confidence in the participants by providing physical activity education and a variety of activities.
  Arms: Intervention

SUMMARY:
Over the past four decades, it has become clear that childhood physical activity carries with it a myriad of beneficial effects. It is closely linked to quality of life and the recognized benefits include, but are not limited to, optimal growth and development, a healthier self-concept, enhanced peer socialization, and decreased anxiety and depression. Long term, an active lifestyle decreases the risk of many important physical and mental morbidities. Thus, the observation that children living with medical conditions and disabilities (MC&D) today, although surviving longer thanks to advances in medical care, are much less active than their peers is a matter of significant concern. Research indicates that the 350,000 Ontario children with MC&D have lower levels of physical activity, higher screen time and more frequent sleep problems.

While the reasons underlying this reality are complex, previous research has identified a substantial subset of children who are motivated to be active but lack the confidence to do so. Fear of pain, concern for MC&D exacerbation and a lack of confidence in individual physical movement capacity contribute to their hesitation. Clinical experience suggests that these children represent 50% to 70% of inactive patients. Research indicates that being motivated to make a change and having the confidence that the desired change can be achieved are the essential precursors upon which successful behaviour change initiatives are built. This randomized, controlled trial will explore whether group sessions with a Registered Kinesiologist lead to a direct bolstering of physical activity confidence, and in turn to increased and sustained physical activity in these children. Such an approach holds the promise of a nonpharmacologic, low cost and accessible means of enhancing health that shall be met with a high level of patient and family support while bringing a significant societal and medical return on investment.

DETAILED DESCRIPTION:
Children living with medical conditions are often unsure about engaging in active play with friends and peers. Some children are worried that physical activity will increase symptoms of their existing illness and increase overall pain. Other children are unable to keep up with peers, or perceive themselves as not good enough to play. This research study will investigate children with medical conditions or disabilities can be supported to become more confident in one' abilities to play actively with their friends. Children who come to our rehabilitation, long term concussion, chronic pain and cardiology clinics will be invited to participate in this project. Children who agree to participate will be assessed three times, in the 1st, 14th and 27th week of the study. During each assessment, children will be asked to complete a short questionnaire about activity preferences and motivation. The child will be given a small activity monitor, about the size of a toonie, which is worn on a belt around the waist. Each child will be asked to wear the monitor for 7 days before returning it to the investigators. After the 1st week of the study, a coin flip will decide the study group for each child. Children in the control group will only do the three assessment visits. Children selected for the exercise group will come to a group physical activity session that will be held once a week for 12 weeks. At each of the 12 sessions, children will be able to try some active games and sports that are suitable for their medical condition or disability. There will be a group of about 8 children, who have similar interests and concerns about physical activity, at each session. The 12 weekly sessions will each be 2.5 hours in length. The study will evaluate how the children's physical activity and confidence to be active change over the 27 weeks, and compare the changes that occur between the children who do or do not attend the 12 weekly physical activity sessions. The results will indicate whether the 12 weekly sessions effectively increase the physical activity confidence of children with medical conditions and disabilities.

ELIGIBILITY:
Inclusion Criteria:

Children with MC&D will be eligible to participate if they meet all of the following criteria:

1. 8 to 17 years of age and actively followed in an out-patient clinic at the Children's Hospital of Eastern Ontario (CHEO);
2. physical activity concerns for the child identified by the patient/parent/healthcare professional;
3. able to participate in physical activity as specified by the responsible physician;
4. a physical disability limiting physical function or concussion symptoms persisting for > 1 month or chronic pain limiting physical function (post physiotherapy treatment) or a cardiac diagnosis;
5. Motivation Ruler score for daily physical activity ≥ 4 (max 10 points) and Confidence Ruler for achieving a change in physical activity < 7 (max 10 points).

Exclusion Criteria:

1. have a cognitive disability that prevents them from completing the study assessments;
2. are unable to complete the assessments or intervention in either English or French;
3. have an acute illness/condition that may impact their physical activity.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Readiness Ruler for Physical Activity Behaviour Change Scores | Baseline, 3 months and 6 months
  Self rating of motivation for physical activity and confidence for making a change in physical activity (both are 1 (low) to 10 (high) scales as per Miller & Rollnick, Motivational Interviewing: Helping People Change, 2012). Eligible patients will have high motivation (> 4/10) but low confidence (< 7/10).
Change in Daily Physical Activity Behaviour | Baseline, 3 months and 6 months
  Actical accelerometer data for 7 day period
Change in Canadian Assessment of Physical Activity Motivation and Confidence Questionnaire Scores | Baseline, 3 months and 6 months
  Valid and reliable assessment of children's motivation and self-confidence for physical activity participation (www.capl-eclp.ca). Maximum score of 10 points, higher score indicates more motivation and confidence.

SECONDARY OUTCOMES:
Change in Screen Time | Baseline, 3 months, and 6 months
  7 day screen time journal
Change in Sleep Time | Baseline, 3 months, and 6 months
  7 day journal

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Longmuir, PhD, Principal Investigator — Children's Hopsital of Eastern Ontario, Research Institute; Hana Alazem, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alazem H, Yaraskavitch J, Blais A, McCormick AM, Lougheed J, Lamontagne C, Goulet KB, Tsampalieros A, Ward LM, Katz SL, Robinson ME, Abbott LS, Kovesi TA, Reisman JJ, Pohl D, Webster RJ, Longmuir PE. Impacting the physical activity confidence of children with medical conditions or disabilities: A randomized controlled trial. Paediatr Child Health. 2025 Mar 27;30(4):257-267. doi: 10.1093/pch/pxae085. eCollection 2025 Jul. PMID 40756554